CLINICAL TRIAL: NCT04149418
Title: Anti-inflammatory Activity of Yogurt Mediated by the Intestine
Brief Title: Yogurt for Prevention of Chronic Inflammation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Wisconsin, Madison (Other)
Collaborators: National Dairy Council (Other); University of Massachusetts, Amherst (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: 2018-1262; A074000 (Other: UW Madison); AG&LSC/FOOD SCIENCE/FOOD SCIEN (Other: UW Madison); Protocol Version 1/10/2019 (Other: UW Madison)
Record Dates: First submitted 2019-10-29; First posted 2019-11-04 (Actual); Last update posted 2022-11-16 (Actual); Status verified 2022-11

CONDITIONS: Obesity; Inflammation
Keywords: yogurt; obesity; intestine
MeSH Terms: conditions — Obesity; Inflammation | interventions — Yogurt; Hazard Analysis and Critical Control Points

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Yogurt-Control (Experimental): Consumption of 12 oz. of low-fat yogurt daily (2 x 6 oz. servings) for 4 weeks, followed by a washout phase for 4 weeks, then consumption of 12 oz. control food (flavored soy pudding, 2 x 6 oz. servings) for 4 weeks.
  Interventions: Other: Yogurt; Other: Control food
- Control-Yogurt (Experimental): Consumption of control food (flavored soy pudding, 2 x 6 oz. servings), followed by a washout phase for 4 weeks, then consumption of 12 oz. of low-fat yogurt daily (2 x 6 oz. servings) for 4 weeks.
  Interventions: Other: Yogurt; Other: Control food

INTERVENTIONS:
Other: Yogurt — Low-fat flavored yogurt
Other: Control food — Low-fat flavored soy pudding

SUMMARY:
The objective of this study is to conduct a randomized cross-over dietary intervention in adult women who are overweight or obese to compare how yogurt and a control food affect biomarkers of inflammation and intestinal health.

ELIGIBILITY:
Inclusion Criteria:

* healthy premenopausal women age 21-55
* BMI ≥ 25 kg/m2
* not taking medication to control hypertension (e.g. anti-hypertensives or diuretics)
* resting blood pressure <140/90 mmHg
* stable body weight for past two months
* willing to maintain a normal exercise level (in general)
* willing to avoid exercise and smoking (or other forms of nicotine intake) for 24 h prior to blood collection
* willing to avoid caffeine for 12 h before study visits
* willing to fast 12 h prior to study visits
* willing to avoid dietary supplements, yogurt and probiotic-containing foods (as necessary) and consume 12 oz. of yogurt and the control food per day (as necessary) for the duration of the study

Exclusion Criteria:

* self-reported previous diagnoses of an inflammatory disease (e.g. inflammatory bowel disease, asthma, arthritis), CVD, diabetes, current cancer treatment (i.e., chemotherapy, radiation therapy)
* have used oral antibiotics in the prior 21 days before sample collection
* actively trying to lose weight
* regularly taking anti-inflammatory drugs
* vegetarian or allergic to soy or dairy
* are pregnant, lactating, or trying to become pregnant

Ages: 21 Years to 55 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Female
Enrollment: 40 (Actual)
Dates: Start 2021-10-15 (Actual); Primary Completion 2022-09-01 (Actual); Study Completion 2022-09-01 (Actual)

PRIMARY OUTCOMES:
Change in Th17 proportion | Baseline, Week 4, Week 8, Week 12
  Change in proportions of circulating Th17 cells (change in control vs. change in yogurt)

SECONDARY OUTCOMES:
Change in Treg proportion | Baseline, Week 4, Week 8, Week 12
  Change in proportion of circulating Treg cells (change in control vs. change in yogurt)
Change in Treg subpopulation | Baseline, Week 4, Week 8, Week 12
  Change in proportion of circulating Treg subpopulation (FoxP3+ IL-10+) (change in control vs. change in yogurt)
Change in Th17 subpopulation (IL-17A+ TNFα+) | Baseline, Week 4, Week 8, Week 12
  Change in proportion of circulating Th17 subpopulation (IL-17A+ TNFα+) (change in control vs. change in yogurt)
Change in Th17 subpopulation (IL-17A+ IFNδ+) | Baseline, Week 4, Week 8, Week 12
  Change in proportion of circulating Th17 subpopulation (IL-17A+ IFNδ+) (change in control vs. change in yogurt)
Change in Th17 subpopulation (IL-17A+ IL-22+) | Baseline, Week 4, Week 8, Week 12
  Change in proportion of circulating Th17 subpopulation (IL-17A+ IL-22+) (change in control vs. change in yogurt)
Change in Th17 subpopulation (IL-17A+ FoxP3+) | Baseline, Week 4, Week 8, Week 12
  Change in proportion of circulating Th17 subpopulation (IL-17A+ FoxP3+) (change in control vs. change in yogurt)
Change in Th17 subpopulation (IL-17A+ IL-10+) | Baseline, Week 4, Week 8, Week 12
  Change in proportion of circulating Th17 subpopulation (IL-17A+ IL-10+) (change in control vs. change in yogurt)
Change in plasma tumor necrosis factor alpha (TNF-alpha) | Baseline, Week 4, Week 8, Week 12
  Change in fasting plasma TNF-alpha (change in control vs. change in yogurt)
Change in plasma interferon gamma (IFN-gamma) | Baseline, Week 4, Week 8, Week 12
  Change in fasting plasma IFN-gamma (change in control vs. change in yogurt)
Change in plasma interleukin-6 (IL-6) | Baseline, Week 4, Week 8, Week 12
  Change in fasting plasma IL-6 (change in control vs. change in yogurt)
Change in plasma interleukin-17A (IL-17A) | Baseline, Week 4, Week 8, Week 12
  Change in fasting plasma IL-17A (change in control vs. change in yogurt)
Change in plasma interleukin-4 | Baseline, Week 4, Week 8, Week 12
  Change in fasting plasma IL-4 (change in control vs. change in yogurt)
Change in plasma interleukin-22 (IL-22) | Baseline, Week 4, Week 8, Week 12
  Change in fasting plasma IL-22 (change in control vs. change in yogurt)
Change in plasma interleukin-10 (IL-10) | Baseline, Week 4, Week 8, Week 12
  Change in fasting plasma IL-10 (change in control vs. change in yogurt)
Change in plasma transforming growth factor beta (TGF-beta) | Baseline, Week 4, Week 8, Week 12
  Change in fasting plasma TGF-beta (change in control vs. change in yogurt)
Change in retinoic acid receptor-related orphan nuclear receptor gamma T (RORgammaT) expression | Baseline, Week 4, Week 8, Week 12
  Change in fasting plasma RORgammaT expression (change in control vs. change in yogurt)
Change in Forkhead box P3 (FoxP3) expression | Baseline, Week 4, Week 8, Week 12
  Change in fasting FoxP3 expression (change in control vs. change in yogurt)
Change in fecal calprotectin | Baseline, Week 4, Week 8, Week 12
  Change in fecal calprotectin (change in control vs. change in yogurt)
Change in fecal tumor necrosis factor alpha (TNF-alpha) | Baseline, Week 4, Week 8, Week 12
  Change in fecal TNF-alpha (change in control vs. change in yogurt)
Change in fecal interleukin 1 alpha (IL-1alpha) | Baseline, Week 4, Week 8, Week 12
  Change in fecal IL-1alpha (change in control vs. change in yogurt)
Change in fecal interleukin 1beta (IL-1beta) | Baseline, Week 4, Week 8, Week 12
  Change in fecal IL-1beta (change in control vs. change in yogurt)
Change in fecal interleukin-6 (IL-6) | Baseline, Week 4, Week 8, Week 12
  Change in fecal IL-6 (change in control vs. change in yogurt)
Change in fecal interleukin-17A (IL-17A) | Baseline, Week 4, Week 8, Week 12
  Change in fecal IL-17A (change in control vs. change in yogurt)

OTHER OUTCOMES:
Change in systolic blood pressure | Baseline, Week 4, Week 8, Week 12
  Change in resting systolic blood pressure (change in control vs. change in yogurt)
Change in diastolic blood pressure | Baseline, Week 4, Week 8, Week 12
  Change in resting diastolic blood pressure (change in control vs. change in yogurt)
Change in BMI | Baseline, Week 4, Week 8, Week 12
  Body mass index (change in control vs. change in yogurt)
Change in Weight | Baseline, Week 4, Week 8, Week 12
  Change in body weight (change in control vs. change in yogurt)
Change in waist circumference | Baseline, Week 4, Week 8, Week 12
  Change in waist circumference (change in control vs. change in yogurt)
Compliance: Number of lids and Unused Containers | Baseline, Week 4, Week 8, Week 12
  Number of lids and unused containers of intervention foods (control vs. yogurt)
Dietary records | 2 Weeks Prior to Intervention, Weeks 0-4, Weeks 4-8, Weeks 8-12
  Comparison of dietary records (control vs. yogurt)
Change in gut microbiota diversity | Baseline, Week 4, Week 8, Week 12
  Change in gut microbiota beta diversity (change in control vs. change in yogurt)
Change in fecal water ex vivo barrier disrupting activity | Baseline, Week 4, Week 8, Week 12
  Change in barrier disrupting activity of fecal water applied to cultured Caco-2 cells (change in control vs. change in yogurt)
Change in fecal total organic carbon | Baseline, Week 4, Week 8, Week 12
  Change in total organic carbon (change in control vs. change in yogurt)
Change in fecal butyrate | Baseline, Week 4, Week 8, Week 12
  Change in fecal butyrate (change in control vs. change in yogurt)
Change in fecal propionate | Baseline, Week 4, Week 8, Week 12
  Change in fecal propionate (change in control vs. change in yogurt)
Change in fecal acetate | Baseline, Week 4, Week 8, Week 12
  Change in fecal acetate (change in control vs. change in yogurt)
Change in fecal bile acid (deoxycholic acid) | Baseline, Week 4, Week 8, Week 12
  Change in fecal deoxycholic acid (change in control vs. change in yogurt)
Change in fecal bile acid (lithocholic acid) | Baseline, Week 4, Week 8, Week 12
  Change in fecal lithocholic acid (change in control vs. change in yogurt)
Change in fecal bile acid (hyodeoxycholic acid) | Baseline, Week 4, Week 8, Week 12
  Change in fecal hyodeoxycholic acid (change in control vs. change in yogurt)
Change in fecal bile acid (3β,12α-Dihydroxy-5β-cholan-24-oic acid) | Baseline, Week 4, Week 8, Week 12
  Change in fecal 3β,12α-Dihydroxy-5β-cholan-24-oic acid (change in control vs. change in yogurt)

CONTACTS AND LOCATIONS:
Overall Officials: Bradley W Bolling, PhD, Principal Investigator — University of Wisconsin, Madison
Locations (1):
- Department of Food Science, Babcock Hall, Madison, Wisconsin, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Hasegawa Y, Noll AL, Lang DJ, Akfaly EM, Liu Z, Bolling BW. Low-fat yogurt consumption maintains biomarkers of immune function relative to nondairy control food in women with elevated BMI: A randomized controlled crossover trial. Nutr Res. 2024 Sep;129:1-13. doi: 10.1016/j.nutres.2024.07.005. Epub 2024 Jul 24. PMID 39153426